CLINICAL TRIAL: NCT05173688
Title: The Relationship Between Different Doses of Propofol and the Occurrence of Dreams in Short Surgery Under General Anesthesia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Shengjing Hospital (Other)
Responsible Party: Principal Investigator, Yanchao Yang, principal investigator, Shengjing Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Propofol and dream
Record Dates: First submitted 2021-11-25; First posted 2021-12-30 (Actual); Last update posted 2022-06-02 (Actual); Status verified 2022-06

CONDITIONS: Dreaming; General Anesthesia
MeSH Terms: interventions — Propofol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Low maintenance dose propofol group (Experimental): The low maintenance dose propofol group was maintained at 4-6 mg/kg/h
  Interventions: Drug: Propofol
- High maintenance dose propofol group (Experimental): The high maintenance dose propofol group was maintained at 8-12 mg/kg/h
  Interventions: Drug: Propofol

INTERVENTIONS:
Drug: Propofol — The low maintenance dose propofol group was maintained at 4-6 mg/kg/h ；and The high maintenance dose propofol group was maintained at 8-12 mg/kg/h

SUMMARY:
Dreams are a remarkable experiment in psychology and neuroscience, conducted every night in every sleeping person. 74% of awakenings from REM sleep resulted in recall of a dream, as compared with only 9% of awakenings from NREM sleep. The association between dreaming and REM sleep was subsequently replicated by many other investigators; typically, around 80% of REM awakenings yield dreams. It became clear over time that there is a good deal of mental activity that occurs during NREM sleep. Typically, it is more thought like, fragmentary, and related to daily concerns than the vivid, hallucinatory, predominantly visual narratives that are most commonly reported from REM sleep. But even this distinction appears not to be absolute. There is now wide acceptance of the view that some dreaming that is indistinguishable from REM sleep dreaming occurs in NREM sleep, most frequently in the sleep-onset period. General anesthesia causes a drug-induced state of unconsciousness and is a non-physiological process that is similar to natural sleep. Patients receiving propofol for maintenance of general anesthesia often report higher incidences of dreaming than patients maintained with volatile anesthetics. One explanation is that propofol and volatile anesthetic have different pharmacological effects in the central nervous system. An alternative explanation is that propofol is associated with more rapid emergence from anesthesia than the older volatile anesthetics, allowing patients to report their dreams before they are forgotten. In order to further verify the hypothesis, the investigators choose gynecological general anesthesia to observe whether the generation of dreams is related to the dose of general anesthesia maintenance .

ELIGIBILITY:
Inclusion Criteria:

* between 18 and 70 years
* with an ASA physical status of I or II

Exclusion Criteria:

* presence of sleep disorders
* pain syndrome
* cardiovascular disease
* sleep apnea syndrome
* psychosis
* history of opioid usage
* history of abnormal operation or anesthesia recovery
* unwillingness to provide informed consent
* a patient with a language communication disorder

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Actual)
Dates: Start 2021-11-30 (Actual); Primary Completion 2022-05-10 (Actual); Study Completion 2022-05-10 (Actual)

PRIMARY OUTCOMES:
Mean blood pressure (systolic and diastolic) | 5 minutes after entering the operation room
  record mean blood pressure during the surgery
Mean blood pressure (systolic and diastolic) | Anesthesia induction to fall asleep
  record mean blood pressure during the surgery
Mean blood pressure (systolic and diastolic) | at the end of surgery
  record mean blood pressure during the surgery
Mean blood pressure (systolic and diastolic) | Upon awakening from anesthesia
  record mean blood pressure during the surgery
Mean blood pressure (systolic and diastolic) | leaving the operation room
  record mean blood pressure during the surgery
heart rate | entering the operation room
  record heart rate during the surgery
heart rate | Anesthesia induction to fall asleep
  record heart rate during the surgery
heart rate | at the end of surgery
  record heart rate during the surgery
heart rate | Upon awakening from anesthesia
  record heart rate during the surgery
heart rate | leaving the operation room
  record heart rate during the surgery
BIS | entering the operation room
  record BIS during the surgery
BIS | Anesthesia induction to fall asleep
  record BIS during the surgery
BIS | at the end of surgery
  record BIS during the surgery
BIS | Upon awakening from anesthesia
  record BIS during the surgery
BIS | leaving the operation room
  record BIS during the surgery
Total dose of propofol | at the end of surgery
  record total dose of propofol
Dream | at the end of surgery
  Dreaming during anesthesia was defined as any experience that was described by the patient as dreaming and was thought by the patient to have occurred between the induction of anesthesia and the first moment of consciousness after anesthesia.27 Awareness was defined as postoperative recall of intraoperative events. All patients who reported dreaming were considered to be "dreamers" for the purpose of the analyses, whether or not they could remember the narrative of the dream. However, only dreaming reports where the narrative was remembered were classified using five-point Likert scales as follows. Emotional content (1 very negative; 5 very positive) ● Memorability (1 can't remember narrative of dream; 5 most memorable ever) ● Visual vividness (1 not at all vivid; 5 most vivid ever) ● Amount of sound (1 no sound; 5 most sound ever)

SECONDARY OUTCOMES:
Postoperative adverse effects | 24 hours after surgery
  record postoperative adverse effects

CONTACTS AND LOCATIONS:
Overall Officials: junchao zhu, Principal Investigator — Shengjing Hospital
Locations (1):
- Shengjing Hospital, Shenyang, Liaoning, China